CLINICAL TRIAL: NCT01521351
Title: A Prospective Natural History Study of Carotid Atherosclerosis
Brief Title: Natural History of Carotid Atherosclerosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Konstantinos Toutouzas, Associate Professor of Cardiology, National and Kapodistrian University of Athens
Other Study IDs: MRcar
Record Dates: First submitted 2012-01-25; First posted 2012-01-30 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Carotid Artery Disease; Stroke; Myocardial Infarction; Angina Pectoris
Keywords: microwave radiometry; cardiovascular events; carotid artery disease; stroke; myocardial infarction
MeSH Terms: conditions — Carotid Artery Diseases; Stroke; Myocardial Infarction; Angina Pectoris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- carotid thermal heterogeneity: Patients that have carotid thermal heterogeneity detected by MR
- no carotid thermal heterogeneity: Patients that DONT have carotid thermal heterogeneity detected by MR
- carotid artery disease: Patients with detected carotid artery disease by ultrasound
- no carotid artery disease: Patients with no carotid artery disease detected by ultrasound

SUMMARY:
A prospective study of 700 patients with coronary artery disease will undergo non invasive evaluation of their carotid arteries by ultrasound and microwave radiometry. The patients will be followed up for 3 years and their outcome regarding the cardiovascular events (death, cardiac events, cerebrovascular events) will be recorded

DETAILED DESCRIPTION:
Carotid artery Thermal heterogeneity recorded by MR will be corelated to cardiovascular events (death, cardiac events, cerebrovascular events) as well as to all demographic (age, sex, hypertension, dyslipidemia, smoking status, etc) factors

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients with coronary artery disease admitted in our hospital

Exclusion Criteria:

* Patients with history of previous cerebrovascular event,
* History of vasculitis, intermittent inflammatory, infectious, or neoplastic conditions likely to be associated with an acute-phase response.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronary artery disease
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2012-01; Primary Completion 2020-06 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
To detect if carotid ultrasound and carotid microwave radiometry measurements can predict the incidence of cerebrovascular and cardiovascular events in patients with coronary artery disease | 3 years
  Microwave radiometry is a non invasive and safe technique that measures temperature of the internal tissues by detecting the normal radiation of the tissues in microwave frequencies. The primary outcome of the study is to see if the temperatures measured in the carotid arteries of patients with coronary artery disease can predict their outcome regarding cerebrovascular and cardiovascular events

SECONDARY OUTCOMES:
Relation of other demographic factors with carotid ultrasound and microwave radiometry measurements and outcome | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos Toutouzas, Principal Investigator — First department of Cardiology, University of Athens Greece
Locations (1):
- First Department of Cardiology, University of Athens, Medical School. Hippocratio Hospital, Athens, Attica, Greece

REFERENCES:
- [Background] Toutouzas K, Grassos H, Synetos A, Drakopoulou M, Tsiamis E, Moldovan C, Agrogiannis G, Patsouris E, Siores E, Stefanadis C. A new non-invasive method for detection of local inflammation in atherosclerotic plaques: experimental application of microwave radiometry. Atherosclerosis. 2011 Mar;215(1):82-9. doi: 10.1016/j.atherosclerosis.2010.12.019. Epub 2010 Dec 23. No abstract available. PMID 21256490
- [Background] Toutouzas K, Benetos G, Drakopoulou M, Deligianni C, Spengos K, Stefanadis C, Siores E, Tousoulis D. Incremental predictive value of carotid inflammation in acute ischemic stroke. Stroke. 2015 Jan;46(1):272-4. doi: 10.1161/STROKEAHA.114.007526. Epub 2014 Nov 4. PMID 25370590
- [Background] Toutouzas K, Benetos G, Drakopoulou M, Bounas P, Tsekoura D, Stathogiannis K, Koutagiar I, Aggeli C, Karanasos A, Panagiotakos D, Siores E, Stefanadis C. Insights from a thermography-based method suggesting higher carotid inflammation in patients with diabetes mellitus and coronary artery disease. Diabetes Metab. 2014 Dec;40(6):431-8. doi: 10.1016/j.diabet.2014.05.005. Epub 2014 Jun 26. PMID 24981292
- [Background] Toutouzas K, Benetos G, Drakopoulou M, Michelongona A, Nikolaou C, Masoura C, Stathogiannis K, Aggeli C, Tsiamis E, Siores E, Stefanadis C. Morphological and functional assessment of carotid plaques have similar predictive accuracy for coronary artery disease. Stroke. 2013 Sep;44(9):2607-9. doi: 10.1161/STROKEAHA.113.002462. Epub 2013 Jul 25. PMID 23887842
- [Derived] Toutouzas K, Benetos G, Oikonomou G, Barampoutis N, Koutagiar I, Galanakos S, Karmpalioti M, Drakopoulou M, Stathogiannis K, Bounas P, Gata V, Antoniadou F, Davlouros P, Alexopoulos D, Hahalis G, Siores E, Sfikakis PP, Tousoulis D. Increase in Carotid Temperature Heterogeneity Is Associated With Cardiovascular and Cerebrovascular Events. Circ Cardiovasc Imaging. 2018 Nov;11(11):e008292. doi: 10.1161/CIRCIMAGING.118.008292. No abstract available. PMID 30571323
- See also: related info — https://scholar.google.gr/citations?user=jksqG1sAAAAJ&hl=el
- See also: Ippocration Hospital — http://www.hippocratio.gr/
- See also: University of Athens Medical School — https://en.uoa.gr/studies/postgraduate_programs/school_of_health_sciences/